CLINICAL TRIAL: NCT05965414
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Pharmacokinetics of Single Ascending Doses and Multiple Ascending Doses of CS6253 in Healthy Volunteers and in APOE4 Carriers
Brief Title: Safety and Pharmacokinetics of Single Ascending Doses and Multiple Ascending Doses of CS6253 in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Artery Therapeutics, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATI-CS-001; 1R44AG076299 (NIH)
Record Dates: First submitted 2023-01-26; First posted 2023-07-28 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Injections

STUDY DESIGN:
Intervention Model Description: SAD:
  5 cohorts 8 of healthy volunteers each will receive single ascending doses of either study drug or placebo (6 active:2 placebo).
  MAD:
  2 or more cohorts 8 of healthy male and female volunteers each will receive single ascending doses of either study drug or placebo (6 active:2 placebo). The subjects will be stratified on their APOE4 status. Each cohort needs to have at least 4 APOE4 carriers.
Who Masked: Participant, Investigator
Masking Description: Neither the investigator nor the subject will know who has received the study drug or the placebo, The injections will be prepared by an unblinded pharmacist according to the randomization list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CS6253 Solution for Injection (Active Comparator): SAD: Single ascending doses: CS6253 Solution for Injection dosing, 50 mg/mL, will be weight based and provided from single use 2 mL vials containing approximately 100 mg CS6253 in phosphate buffered saline (PBS) solution
  MAD: Multiple ascending doses (4x every 72 hours): CS6253 Solution for Injection dosing, 50 mg/mL, will be weight based and provided from single use 2 mL vials containing approximately 100 mg CS6253 in phosphate buffered saline (PBS) solution
  Interventions: Drug: CS6253 Solution for Injection
- Placebo (Placebo Comparator): SAD and MAD: Placebo control will be provided from vials containing physiological saline for injection in an equal amount as necessary for the active arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CS6253 Solution for Injection — Solution for intra-venous injection, 50mg CS6253 /mL. Single-use vials containing 100 mg CS6253 (2 mL of 50 mg/mL concentration)
  Arms: CS6253 Solution for Injection
Drug: Placebo — Physiological saline solution for intra-venous injection
  Arms: Placebo

SUMMARY:
* Phase 1A SAD: Five or more cohorts of 8 healthy volunteers (HVs) will receive a single IV bolus injection of study drug or placebo. The first 4 cohorts will be male only. The last cohort will be repeated with the max safe dose of the previous cohorts in healthy elderly subjects (male and female of non childbearing potential, > 50years)
* Phase 1B MAD: Two or more cohorts of 8 male and female HVs will receive multiple (4) IV bolus injections of study drug or placebo every 72 hours.
* Phase 1 Subcutaneous SC Cohort: One cohort of 6 male and 6 female HVs will receive one SC injection of study drug.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study in HV and in APOE4 carriers.

Phase 1A Single Ascending Dose (SAD): In 5 or more sequential SAD cohorts of 8 (6 active:2 placebo) HVs a single IV bolus injection (CS6253 1, 2.4, 6, and 10 mg/kg or placebo) will be administered and PK, safety, and biomarkers will be assessed. The first 4 cohorts will include males only. In the fifth cohort 8 (6 active:2 placebo) subjects, male and female of non-childbearing potential and at least 50 years old, will be administered CS6253 at equal to or lower doses than the maximum safe SAD dose in HV.

CSF will not be collected in the first 2 SAD cohorts. In the following cohorts, CSF will be collected before dosing and over 24 hours after dosing. Additional cohorts may be added as needed and deemed safe and appropriate by the Data Safety Monitoring Board (DSMB).

Phase 1B Multiple Ascending Dose (MAD): In 2 or more sequential MAD cohorts of 8 (6 active:2 placebo) male and female HVs at least 50 years old on average ≥ 3/sex/cohort; ≥ 4 APOE4 carriers/cohort, will be administered multiple IV bolus injections. Cohort 1 will be administered CS6253 at 75% of the maximum safe SAD dose in subjects at least 50 years old or placebo, and if no Treatment Emerging Adverse Events (TEAEs), in Cohort 2 at 100% of the maximum safe SAD dose or placebo will be administered every 72 hours x 4 doses and PK, safety, and biomarkers will be assessed. Plasma PK will be assessed after first and fourth dose in all cohorts. CSF will be collected before dosing and over 24 hours in conjunction with the fourth dose. Cohorts of 8 subjects (6 active:2 placebo) may be added at doses equal to or lower than the maximum safe MAD dose to further explore CS6253 brain exposure and Pharmacodynamics (PD) dependency on APOE4 isoform and sex.

Phase 1 Subcutaneous SC Cohort: One cohort of 6 (>=4) male and 6 (>=4) female HVs will receive one SC injection of study drug. From these 12 subjects (>=4) female and (>=4) male subjects need to be an APOE4 carrier.

ELIGIBILITY:
Inclusion Criteria:

1. Male HVs at least 18 years old.
2. a) Cohort 5 only: Male and female HVs at least 50 years old and if female be of non-childbearing potential, i.e. meet at least one of the following criteria: postsurgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or postmenopausal (amenorrheic for at least 2 years and a serum follicle-stimulating hormone (FSH) > 30 IU/L).

   b) If subject is male, must be willing to use acceptable contraception from Day 1 until 30 days after the last dose of study drug.
3. The subject has a body mass index (BMI) within 18-32 kg/m² (inclusive).
4. The subject is in reasonably good health as determined by medical history and physical examination and clinical laboratory tests.
5. The subject is willing and able to speak, read, and understand Spanish and give signed informed consent.
6. The subject must agree to comply with a lumbar catheterization and collection of blood and CSF samples (SAD Cohorts 3-5 only and MAD cohorts).
7. The subject is willing and able to comply with all testing and requirements defined in the protocol.
8. The subject is willing, deemed compliant, and able to remain at the Clinical Research Unit (CRU) for the duration of the confinement period and return for all outpatient visits.

Phase 1B MAD

The eligibility criteria for the Phase 1B MAD study are the same as described for Phase 1A SAD, with the following exceptions:

1. At least 50 years old and female need to be of non-childbearing potential
2. Known to have at least 1 APOE4 allele (homozygous or heterozygous). Note: this criterion applies to on average for the MAD at least 4 APOE4 subjects per cohort.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled:

1. The subject has any clinically significant deviations from normal in physical examination, ECG, or clinical laboratory tests, as determined by the investigator.
2. The subject has an increased bleeding risk or is treated with anti-coagulation therapies including but not limited to aspirin, coumarin, warfarin and heparin.
3. The subject has had a clinically significant illness within 30 days of check-in, as determined by the investigator.
4. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
5. History of Type 2 diabetes mellitus or hemoglobin A1c (HbA1c) > 7%.
6. Fasting triglycerides > 400 mg/dL
7. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 (Cockcroft-Gault formula)
8. The subject has changed the frequency or dose of chronic medication within the last 8 weeks.
9. The subject has a history of substance abuse or a positive alcohol or urine drug screen at screening or at check-in.
10. The subject has a positive serum hepatitis B surface antigen or positive anti-hepatitis C virus test at the Screening Visit.
11. Have positive test results for, or evidence of active infection with, human immunodeficiency virus type 1 or 2, or hepatitis B, or C.
12. The subject has received an investigational drug within 30 days of Check-in.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CS6253 | SAD: After dosing and until 72 hours after dosing; MAD: After dosing until day 13 (72 hours after the last dosing on day 10)
  All treatment emerging Adverse Events (TAEs) will be recorded until the SAD: Day 4 and MAD: Day 13
SAD-Plasma: AUC0-last | Pharmacokinetics (PK) samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Area under the concentration-time curve until the last quantifiable concentration
SAD-Plasma: AUC0-inf | PK samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Area under the concentration time curve from time 0 extrapolated to infinity
SAD-Plasma: Cmax | PK samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Maximum observed plasma concentration (eg C0)
SAD-Plasma: Kel | PK samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Terminal elimination rate constant
SAD-Plasma: t1/2 | PK samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Terminal elimination half-life
SAD-Plasma: Clearance (CL/F) | PK samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Apparent clearance
SAD-Plasma: Vd/F | PK samples will be collected at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48, and 72 hours postdose; MAD:
  Apparent volume of distribution
SAD-Cerebrospinal Fluid (CSF): AUC0-last | PK samples will be collected by lumbar catheter starting predose, and at 0.5, 2, 8, 12 and 24 hours postdose.
  In cohorts 3-5:Area under the concentration-time curve in CSF until the last quantifiable concentration
SAD-CSF: Cmax | PK samples will be collected by lumbar catheter starting predose, and at 0.5, 2, 8, 12 and 24 hours postdose.
  In cohorts 3-5:Maximum observed CSF concentration (eg C0)concentration
MAD-Plasma: AUC0-last | PK samples will be collected after the first and fourth doses (Day 1 and Day 10) at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72 hours postdose.
  Area under the concentration-time curve until the last quantifiable concentration
MAD-Plasma: Cmax | PK samples will be collected after the first and fourth doses (Day 1 and Day 10) at predose and at 0.16, 0.5, 1, 2, 4, 8, 12, 24, 48 and 72 hours postdose.
  Maximum observed plasma concentration (eg C0)
MAD-CSF:AUC0-last | CSF collection by lumbar puncture (LP) will be performed before the first dose. At the fourth dose, on Day 10, serial CSF samples will be collected by lumbar catheter starting predose, and at 0.5, 2, 8, 12 and 24 hours postdose.
  Area under the concentration-time curve until the last quantifiable concentration
MAD-CSF: Cmax | CSF collection by lumbar puncture (LP) will be performed before the first dose. At the fourth dose, on Day 10, serial CSF samples will be collected by lumbar catheter starting predose, and at 0.5, 2, 8, 12 and 24 hours postdose.
  Maximum observed CSF concentration (eg C0)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M. Borobia Perez, MD, Ass.Prof, Principal Investigator — Universidad Autónoma de Madrid, Farmacología y Terapéutica / Facultad de Medicina
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared